CLINICAL TRIAL: NCT06768385
Title: Comparison of The Efficacy of TAP and TAPA (Thoracoabdominal Nerve Blockage With Perichondrial Approach) Blocks For Pain Treatment After Laparoscopic Cholecystectomy
Brief Title: Comparison of Two Regional Blocks For Pain Treatment After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Dilek Yamac, MD, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBU-ANESTHESİA-DMY-02
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Pain, Postoperative
Keywords: laparoscopic cholecystectomy; transversus abdominis plane block; thoracoabdominal nerve block with the perichondral approach
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion; tapasin

STUDY DESIGN:
Intervention Model Description: The patients were randomly allocated to one of two groups using a computer-generated randomized sequence table with an allocation ratio of 1:1 and a block size of two.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study was conducted using a sealed envelope system. The sealed, opaque, sequentially numbered envelopes were opened by intervention staff who conducted induction of anesthesia and block procedure just prior to surgery. A second investigator involved in the assessment of postoperative outcomes and another investigator involved in data collection were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group T (Active Comparator): After general anesthesia induction, TAP block was applied to Group T. TAP block is the application of local anaesthetic agents to the neurofascial space between the internal oblique and transversus abdominis muscle layers located in the anterolateral region of the abdomen.
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- group P (Active Comparator): TAPA block was applied to Group P. In TAPA block, local anesthesia is applied to two points, the upper part of the chondrium and the lower part of the chondrium.
  Interventions: Procedure: thoracoabdominal nerve blockage with perichondrial approach (TAPA) block

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block — : It was performed under USG guidance using 30 ml of 0.25% bupivacaine with an 80 mm insulated peripheral block needle. Local anaesthetic was applied between the upper fascia of the transversus abdominus muscle and the fascia of the internal oblique muscle at the midpoint of the distance between the costal margin and the iliac crest in the midaxillary line under USG imaging guidance.
  Arms: group T
Procedure: thoracoabdominal nerve blockage with perichondrial approach (TAPA) block — Under USG guidance, 20 ml of 0.25% bupivacaine was administered between the upper fascia of the transversus abdominis muscle and the lower fascia of the costochondral tissue at the level of the 9th and 10th ribs (arcus costarum) in the midclavicular line with an 80 mm insulated peripheral block needle. Then, 10 ml of 0.25% bupivacaine was injected into the upper fascia of the costochondral tissue and the lower fascia of the external oblique muscle. The block was performed by following the needle path in the ultrasound image.
  Arms: group P

SUMMARY:
In laparoscopic cholecystectomies, ultrasound-guided interfascial plane blocks are commonly used for postoperative analgesia. The aim of our study was to compare the postoperative analgesic efficacy of thoracoabdominal nerve block with the perichondral approach (TAPA) with transversus abdominis plane (TAP) block in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is one of the most frequently performed surgical operations and the postoperative hospital stay is short (1). Although there is less postoperative pain in laparoscopic surgeries than in open surgeries, severe pain is a common complaint, especially in the first 24 hours. Therefore, various modalities have been tried to reduce postoperative pain (2).

In recent years, the effectiveness of ultrasound-guided interfascial plane blocks has come to the fore in the field of regional anaesthesia and pain management. There has always been a search for a regional anaesthesia method that provides effective analgesia of the anterolateral part of the upper abdomen. In addition to anterolateral blocks, such as pectoralis nerve block (PECS) and serratus intercostal plane block (SIBP), other posterior blocks like quadratus lumborum blocks and erector spinus plane blocks have been used for this purpose. TAP block is the application of local anaesthetic agents into the neurofascial space between the internal oblique and transversus abdominis muscle layers located in the anterolateral region of the abdomen. This procedure, in which the anterior branches of the 7th-12th thoracic intercostal and first lumbar (L1) nerves are blocked, is frequently used to provide pain control after operations involving the abdominal and inguinal regions (3,4).

Recently introduced thoracoabdominal nerve blockage with perichondrial approach (TAPA) has been reported to provide sensory blockade between midaxillary line and midabdominal/sternum in dermatomes between T5-T12 (5,6). In TAPA block, local anesthesia is applied to two points, the upper part of the chondrium and the lower part of the chondrium. In this way the anterior and lateral cutaneous branches of the intercostal nerves are blocked. In light of this information, our hypothesis is that the analgesic effect will be greater in TAPA block since the lateral branches of the intercostal nerves are also affected.

The aim of our study is to compare the postoperative analgesic efficacies of TAP and TAPA blocks to be applied to patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:Patients classified as I-II-III by the American Society of Anesthesiologists (ASA) and aged between 20 and 70 years were included in the study

Exclusion Criteria:Patients were excluded if they were younger than 20 years, older than 70 years, had ASA physical status classification IV, were pregnant or had a body mass index (BMI) ≥ 35 kg m-2, had a skin infection at the needle puncture site, had a history of previous abdominal surgery or trauma, were known to be allergic to any of the study drugs, had used any analgesic within 24 hours before surgery, had a history of chronic opioid use, alcohol or drug use, were receiving antithrombotic therapy, and had abnormal coagulation parameters.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative analgesic efficacy | At the postoperative 2nd, 6th, 12th and 24th hours, the patient's request and administrations from the patient-controlled analgesia (PCA) device, total tramadol dose and the first additional analgesic drug if needed, and application times were recorded.
  NRS (Numerical Rating Scale) was used for pain monitoring. Patients were informed about the NRS assessment for pain. It was stated that a score of 0 meant no pain and a score of 10 meant the worst pain imaginable. After the first assessment hour when NRS >4 was noted in patients, IV analgesia treatment was started (dexketoprofen 50 mg IV as additional analgesic). If NRS <4 and the patient did not request analgesic, the drug dose was skipped.

SECONDARY OUTCOMES:
presence of nausea-vomiting | the postoperative 2nd, 6th, 12th and 24th hours
  presence of nausea-vomiting recorded at the postoperative 2nd, 6th, 12th and 24th hours

CONTACTS AND LOCATIONS:
Overall Officials: Dilek M Yamac, Principal Investigator — Sultan Abdülhamid Han education and research hospital
Locations (1):
- SBU Sultan Abdulhamid Han, Istanbul, Asia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No